CLINICAL TRIAL: NCT05810519
Title: The Effect of an Active Break Intervention on Nonspecific Low Back Pain and Musculoskeletal Discomfort During Prolonged Sitting Among Young People (SPINE-have&Care)
Brief Title: Active Break Intervention on Low Back Pain and Musculoskeletal Discomfort During Prolonged Sitting Among Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Collaborators: University of Tehran (Other)
Responsible Party: Principal Investigator, Magdalena Plandowska, PhD, Józef Piłsudski University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3/BN/UPB/2023
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain
Keywords: non-specific low back pain; young people; sitting position; break; active break
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants assigned to the experimental group will receive recommendation to take an active break with the proposed lumbar and hip extension exercises for every 30 minutes of sitting.
  Interventions: Behavioral: Active break with the proposed lumbar and hip extension exercises
- Control group (Active Comparator): Participants assigned to the control group will receive an self-care recommendations book.
  Interventions: Behavioral: Self-care recommendations

INTERVENTIONS:
Behavioral: Active break with the proposed lumbar and hip extension exercises — Participants assigned to the experimental group will receive recommendation to take an active break with the proposed lumbar and hip extension exercises for every 30 minutes of sitting. In the experimental intervention, the exercise program include exercises and will be based on patient education. The participants will also explain the importance of regular training and receive a booklet with photographed and described exercises.
  Arms: Experimental group
Behavioral: Self-care recommendations — Participants assigned to the control group will receive an educational self-care book containing information on low back pain, anatomy of the spine and its relation to the muscular chain, care during daily life activities and the importance of regular physical exercises. The control group will perform their regular baseline activities.
  Arms: Control group

SUMMARY:
The most recent evidence showed that the COVID-19 (coronavirus disease 2019, National Institutes of Health) pandemic caused an increase in low back pain (LBP) prevalence and intensity among young people. This may be explained by the prolonged sitting time, next to reduced level of physical activity. Young people spend most of their time in a sitting position while studying (in school class, during homework) and using electronic devices (using the computer, laptop, mobile phone, tablets, or watching TV), and now using e-learning methods. E-learning, and thus prolonged sitting, is a topic that returned to higher education at the beginning of the 2022-2023 academic year because of the current energy crisis. Re-education on sitting posture is a common aspect of LBP management. Physiotherapists recommend many different sitting positions to prevent and treat the negative effects of prolonged sitting. However, there is debate regarding what is an optimal sitting posture. Studies showed that sitting posture with the backrest on the chair induced minimal changes in lumbar lordosis and significantly lesser pain compared to other types of the chair. Even though the sitting posture will be followed by proper ergonomic principles, every position (lordotic or kyphotic) maintained for a prolonged time leads to discomfort and soft tissue symptoms. Studies showed that body perceived discomfort scores increased over time during sitting and after 30 min of sitting is significantly greater than those at baseline. Currently, breaks are recommended for mitigating the adverse of prolonged sitting, but more evidence is needed to verify effectiveness of breaks. The aim of this study is to evaluate the effect of active break on reduce LBP and perceived musculoskeletal discomfort during prolonged sitting in young people with LBP. Optimal combination of sitting and breaks will help to develop ergonomic recommendations for young people. Main research outcomes - exercise protocol and intervention - will be developed to match the needs of young people with LBP and the possibilities of the environment, in order to reduce LBP and musculoskeletal discomfort during prolonged sitting, and consequently, maintain health and quality of life. The intervention will address the social and health needs of a particular social group: young people, with the possibility of extending the recommendations to other groups.

DETAILED DESCRIPTION:
Background:

Young people tend to spend most of their time in sitting position while studying (in the school class, during homework) and using the electronic devices (using the computer, laptop, mobile phone, tablets or watching TV). Moreover, during the COVID-19 (coronavirus disease 2019, National Institutes of Health) pandemic, many countries switched their teaching programs into e-learning, where students spend long hour using electronic devices. Now e-learning methods have been often used, not only during pandemic. The current energy crisis, exacerbated by the war in Ukraine, is causing e-learning back to educational institutions. However this change in learning methods is associated with musculoskeletal dysfunction including low back pain (LBP). Low back pain was one of the most common musculoskeletal disorders and today it is known that the COVID-19 pandemic has increased the prevalence and intensity of LBP. This may be explained by the prolonged sitting time, next to reduced level of physical activity. Most people sit for a long hours in a slumped sitting posture. Prolonged sitting causes changes in the passive structures of the spine and induces a low back compressive load significantly higher than that observed in standing. Physiotherapists recommend many different sitting positions to prevent and treat negative effects of prolonged sitting. However, there is debate regarding what is an optimal sitting posture. Periodic rest breaks have been identified as a way to reduce self-report discomfort at the low back and a standing breaks may be beneficial for the passive tissues of the spine. A combination of sitting and standing is beneficial for reducing musculoskeletal discomfort.

Research aim:

The aim of this study is to evaluate the effect of active break on reduce LBP and perceived musculoskeletal discomfort during prolonged sitting in young people with LBP.

Methods:

This will be a randomized controlled study with pre and post-intervention assessment. The participants will be recruited from students. Participants were randomly assigned to the intervention group consisting of an active break (n = 25) or the control group (n = 25). The group with an active break with postural change from sitting to standing will be recommended to take an active break for every 30 minutes of sitting. The primary outcome will be average pain intensity (Visual Analogue Scale, VAS), disability measured using the Oswestry Disability Index and perceived musculoskeletal discomfort during prolonged sitting (Borg scale) and The Global Perceived Effect (7-point Likert scale). Secondary outcome will Post-Intervention Questionnaire (5-item self-completed questionnaire).

Expected outcomes:

Research outcomes - exercise protocol and intervention - will be developed to match the needs of young people with LBP and the possibilities of the environment, in order to reduce LBP and musculoskeletal discomfort during prolonged sitting, and consequently, maintain health and quality of life. The intervention will address the social and health needs of a particular social group: young people, with the possibility of extending the recommendations to other groups. Research outcomes will build evidence-based practice for students, teachers, health professionals, personal trainers, and family doctors.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 25 years of age;
* participants with non-specific low back pain (defined as pain and discomfort localized below the costal margin and above the inferior gluteal folds), pain of at least 3 months' duration, without radiation to legs;
* participants who did not have a surgical history due to spinal problems;
* participants who did not have radiculopathy or other injuries such as fractures, stenosis or tumors in the spine;
* participants who had not received any treatment related to low back within the last six months;
* participants who had not used medication for low back pain in the last three months.

Exclusion Criteria:

* spinal pathology (eg, tumor, infection, fracture, inflammatory disease),
* patients with disc herniation and leg length discrepancy;
* pregnancy,
* nerve root compromise,
* previous spinal surgery,
* major surgery scheduled during treatment or follow-up period,
* presence of any contraindication to exercise.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Change from Pre-Intervention (baseline) compared to Post-Intervention (12 weeks)
  Pain will be measured through Visual Analogue Scale (VAS, in centimeters). 0 represents "no pain" and 10 "worst pain possible".
Disability | Change from Pre-Intervention (baseline) compared to Post-Intervention (12 weeks)
  Level of functional disabilities of participants resulting from LBP would be measured using Revised Oswestry Low Back Pain Disability Index
Perceived musculoskeletal discomfort during prolonged sitting | Change from Pre-Intervention (baseline) compared to Post-Intervention (12 weeks)
  Perceived musculoskeletal discomfort during prolonged sitting will be measured using the Borg CR-10 scale during the 1 hour of sitting. Participants will indicate which parts of their body experienced musculoskeletal discomfort and how much discomfort was felt (on a scale of 0-10; 0 denotes no discomfort and 10 denotes extreme discomfort).
The Global Perceived Effect | Completion of 12 week intervention
  The global perceived improvement will be assessed using The Global Perceived Effect Scale (GPE, 7-point numerical scale). The participants will be asked: 'Since the start of treatment, my current overall status is: 1 = completely recovered, 2 = much improved, 3 = slightly improved, 4 = not changed, 5 = slightly worsened, 6 = much worsened and 7 = worse than ever. These ratings will be dichotomized into "improved" (GPE scores 1-2) and "not improved" (GPE scores 3 to 7).

SECONDARY OUTCOMES:
Post-Intervention Questionnaire | Completion of 12 week intervention
  The postIQ will be focused on the subjective opinions of the participants in relation to the Active Break Program. The items will be presented in the form of statements to which students will be asked to respond using a 1-5 Likert scale ("strongly agree", "agree", "not sure", "disagree", and strongly disagree").

CONTACTS AND LOCATIONS:
Locations (1):
- Jozef Pilsudski University of Physical Education in Warsaw, Faculty of Physical Education and Heath in Biala Podlaska, Biała Podlaska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plandowska M, Labecka MK, Truszczynska-Baszak A, Plaszewski M, Rajabi R, Makaruk B, Rozanska D. The Effect of an Active Break Intervention on Nonspecific Low Back Pain and Musculoskeletal Discomfort during Prolonged Sitting among Young People-Protocol for a Randomized Controlled Trial. J Clin Med. 2024 Jan 22;13(2):612. doi: 10.3390/jcm13020612. PMID 38276118
- [Derived] Labecka MK, Plandowska M, Truszczynska-Baszak A, Rajabi R, Rozanska D, Plaszewski M. Effects of the active break intervention on nonspecific low back pain among young people: a randomized controlled trial. BMC Musculoskelet Disord. 2024 Dec 20;25(1):1055. doi: 10.1186/s12891-024-08186-3. PMID 39707287